CLINICAL TRIAL: NCT04740853
Title: Investigation of the Effectiveness of Sensory Integration Therapy in Children With Dyslexia
Brief Title: Sensory Integration Therapy in Children With Dyslexia
Acronym: Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Remziye Akarsu, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rakarsu
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Dyslexia
Keywords: Dyslexia, sensory integration therapy, MOHO.
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Integration Therapy+Special Education (Experimental): The therapy program was prepared and applied according to the Ayres theory and based on the basic principles of sensory integration therapy prepared by Parham depending on the evaluation results. Therapy was applied to the intervention group, with a 45-minute session+15 minutes of family information once a week for eight weeks, in addition to the special education sessions they received twice a week in special education institutions. The sensory integration therapy included sensory diet practices and activities consisting of vestibular, tactile, proprioceptive, auditory and visual stimuli.
  The intervention group continued special education sessions in special education and rehabilitation centers twice a week for eight weeks. In the special education sessions, reading, writing, sequencing, arithmetic, language, organization, memory studies were applied.
  Interventions: Behavioral: Sensory Integration Therapy+Special Education
- Special Education (Active Comparator): The control group continued special education sessions in special education and rehabilitation centers twice a week for eight weeks. Within the scope of special education sessions, reading, writing, sequencing, arithmetic, language, organization, memory studies were applied.
  Interventions: Behavioral: Sensory Integration Therapy+Special Education

INTERVENTIONS:
Behavioral: Sensory Integration Therapy+Special Education — Sensory integration is a theory first put forward by Ayres in 1972. It is a neurological process that organizes sensory stimuli from our body and our environment for use in the daily life. When the sensory integrity organization of individuals is provided, it is possible to use their body effectively against the environment. Sensory integration therapy, which is defined as a physiologically based process by Ayres and Dunn, also provides changes in individuals' occupations.

SUMMARY:
The aim of this study is to examine the sensory and functional effects of sensory integration therapy in children with dyslexia according to the Model of Human Occupation (MOHO).

35 participant (17 intervention, 18 control, aged 8.7;8.5 years) diagnosed with dyslexia were included in the study. In the special education and rehabilitation centers, where they were followed, both groups received special individual training sessions twice a week for eight weeks, and in addition to the intervention group, sensory integration therapy was applied once a week for eight weeks (45 minutes therapy, 15 minutes family briefing - 60 minutes in total). Sensory Profile Test was used for sensory processing evaluation and SCOPE (The Short Child Occupational Profile) for occupational performance analysis. Intervention results and intergroup scores were analyzed using the Wilcoxon Paired Two Sample Test and the Mann Whitney-U test.

DETAILED DESCRIPTION:
This study aims to examine the effect of sensory integration therapy on sensory modulation and daily functional performance in children with dyslexia, according to the occupational therapy model MOHO.

The study was carried out in Biruni University Sensory Integration Unit on 35 participants ( intervention group:17, aged 8,7±0,85 years; control group:18, aged 8,5±1,1 years) with dyslexia.

According to the results of the analysis made in the R program, it was calculated that the sample volume should be 35 at 80% Power.

The investigators talked about the study with a special education and rehabilitation center. They will briefly ask the families of children with dyslexia who meet the inclusion criteria, during their routine education/therapy sessions, whether they might be interested in taking part in the study or not. Following this, the informed consent form was signed by the parents who accepted and were willing to volunteer to take part in the study, since the individuals participating in the study were under the age of 18.

Children between the ages of 6 and 10 years who were diagnosed with dyslexia by a psychiatrist according to DSM-V criteria were included in the study. Children with any secondary diagnosis were excluded from the study. 40 participants were randomly divided into 20 control and 20 intervention groups using a random number table.

Children in the intervention group were included in sensory integration therapy sessions at Biruni University Sensory Integration Unit for eight weeks, one session a week, 45 minutes sessions, and 15 minutes of family information. Both groups continued special education sessions in special education and rehabilitation centers twice a week for eight weeks. Three participants from the intervention group and two participants from the control group left the study.

The socio-demographic data was collected and recorded, including age, parentage, gender, health status. During the evaluation phase, the Sensory Profile test and the SCOPE (The Short Child Occupational Profile) was applied to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Were between the ages of 6 and 10 years
* Diagnosed with dyslexia by a psychiatrist according to DSM-V criteria

Exclusion Criteria:

• Had any secondary diagnosis

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The Sensory Profile Test | 2 weeks
  The Sensory Profile Test is an assessment tool for sensory modulation developed by Winnie Dunn and it is used to determine the types of sensory response during daily activities and which sensory systems are most affected. Functional performance is a valid and reliable assessment tool for measuring sensory processing skills. In the scale, there are 125 questions asked to parents, divided into three parts as sensory processing, modulation, and behavioral-emotional responses. It is evaluated according to the Likert scale (1 = Always, 2 = Frequently, 3 = Sometimes, 4 = Rarely, 5 = Never) with 9 factor scores consisting of these parameters. Typical performance, probably difference and definite difference score ranges are determined for each parameter. Total score for each parameter; There is an improvement from the absolute difference score range to the typical performance score range.
The Short Child Occupational Profile | 2 weeks
  The SCOPE is an assessment tool to evaluate children's activity participation within the framework of MOHO. This questionnaire consists 25 questions (4 questions from each performance area of MOHO and 5 questions for the environment) and it is scored 4-point likert scale. The higher scores mean better performance. The SCOPE is a scale with proven validity and reliability, in which activities, roles and tasks are evaluated comprehensively, the child's skills and environmental opportunities are examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Remziye Akarsu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No